CLINICAL TRIAL: NCT05244044
Title: Changes in Functional Exercise Capacity After PUlmonary REhabilitation in Primary Care: a Randomized, Controlled, Multicenter, Pragmatic Trial in 134 Patients With Long COVID (PuRe-COVID)
Brief Title: Pulmonary Rehabilitation for Long COVID (Post COVID-19 Condition)
Acronym: PuRe-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other); Universiteit Antwerpen (Other); Hasselt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UZA
Record Dates: First submitted 2022-02-14; First posted 2022-02-17 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-05

CONDITIONS: COVID-19; Long COVID; Post COVID-19 Condition
Keywords: Pulmonary rehabilitation; Physiotherapy; Respiratory physiotherapy
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Primary Health Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessor of the 6MWT (the primary outcome) is blinded. Also the assessor of the lung function, MIP/MEP and hand grip strength is blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary rehabilitation group (Active Comparator): The intervention group receives a 12 weeks pulmonary rehabilitation program supervised by a primary care physiotherapist consisting of maximum 36 sessions (3 sessions per week).
  Interventions: Other: Pulmonary rehabilitation in primary care
- Control group without rehabilitation (No Intervention): The control group will receive usual care that doesn't include pulmonary rehabilitation or a supervised physical activity program.

INTERVENTIONS:
Other: Pulmonary rehabilitation in primary care — Pulmonary rehabilitation consists breathing exercises, exercise capacity, muscle strength and change towards an active lifestyle.
  Arms: Pulmonary rehabilitation group

SUMMARY:
In the PuRe COVID study (a randomized, controlled, multicenter, pragmatic trial) the investigators aim to assess the effect of a pulmonary rehabilitation program in primary care on exercise capacity (6MWT) and daily life physical activity in patients with long COVID.

134 patients with long COVID, defined by self-reported persistent COVID related symptoms ≥6 weeks after COVID-19 infection and a positive symptom score (CAT score ≥10 or mMRC score ≥2 or CIS-fatigue ≥36 or PCFS score of ≥2), will be recruited and divided into an intervention group or a control group. The intervention group will get twelve weeks of primary care pulmonary rehabilitation (PR) including coaching by primary care physiotherapists. The control group consists of usual care, which does not include a pulmonary rehabilitation program.

This study will help determine whether the type of symptoms or affected body system can impact recovery form long covid during rehabilitation and after follow-up. The investigators will analyze determinants and risk factors that characterize non-responders and non-adherers to better understand which patients with long COVID benefit from rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with status post COVID-19 (positive COVID-19 PCR or an official pharmacy performed antigen test or a self-performed test confirmed by a physician during the acute COVID-19 ≥ 6 weeks ago or positive antibodies before vaccination or positive antibodies before vaccination).
* Persistent COVID related symptoms that were not present pre-COVID-19 or were less severe pre-COVID.
* Symptomatic: quantified by dyspnea on exertion, loss of energy, fatigue or sleep impairment based upon the score of four questionnaires:

  * COPD Assessment Test (CAT) ≥10, and/or
  * modified Medical Research Council dyspnea scale (mMRC) ≥2, and/or
  * CIS-fatigue ≥36, and/or
  * post-COVID-19 Functional Status (PCFS) ≥2.

Exclusion Criteria:

* Patients with known or self-reported cognitive, hearing, visual, neurological or musculoskeletal conditions that make it impossible to participate in pulmonary rehabilitation.
* Prior physiotherapy for long COVID if:

  * patients who have completed ≥9 sessions of physiotherapy in total for long COVID.
  * patients who completed any physiotherapy session in the previous 12 weeks for long COVID (primary care or hospital based; pulmonary or non-pulmonary).
* Patients with predominantly neurological disorders impacting respiratory function will not be eligible for the study.
* Patients that are not able to give informed consent or not able to complete questionnaires.
* Patients who have had any organ transplatation in the past, have to undergo any transplantation or are on an active transplantation list.
* Patients with active malignancy and/or (maintenance) treatment for active malignancy or curatively treated carcinoma within the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Exercise capacity | Baseline - 12 weeks
  Change in functional exercise capacity measured by 6-minute walk test (6MWT).

SECONDARY OUTCOMES:
Change in physical activity | Baseline - 12 weeks
  Change in physical activity as objectively measured by an activity tracker (number of steps).
Change in COVID-19 related symptoms | Baseline - 12 weeks - 24 weeks - 36 weeks
  The COVID-19 related symptoms will be measured with the COPD assessment test (CAT). The total CAT score ranges from 0 to 40 where 0 represents no symptoms and 40 very bad symptoms.
Change in quality of life | Baseline - 12 weeks - 24 weeks - 36 weeks
  The quality of life will be measured with the EQ-5D-5L.
Change in fatigue | Baseline - 12 weeks - 24 weeks - 36 weeks
  The changes of the level of fatigue will be measured with the Checklist Individual Strength -fatigue (CIS-fatigue) score. The total CIS-fatigue score ranges from 20 to 140 where 20 represents no symptoms and 140 very bad symptoms.
Change in dyspnoea | Baseline - 24 weeks - 36 weeks
  Changes in dyspnoea, measured with the modified medical research council (mMRC). The total mMRC scale ranges from 0 to 4 score where 0 represents no dyspnoea and 4 a lot of dyspnoea.
Change in functional status | Baseline - 12 weeks - 24 weeks - 36 weeks
  The functional status will be measured by the post COVID-19 functional status scale (PCFS). It is an ordinal score ranging from 0 to 4 where 4 means the patient has a lot of limitations in daily life.
Change in work productivity and activity impairment. | Baseline - 24 weeks - 36 weeks
  This will be measured with the "work productivity and activity impairment" questionnaire (WPAI), consisting of 6 questions.
Change in anxiety and depression symptoms. | Baseline - 24 weeks - 36 weeks
  This will be measured by the Hospital Anxiety and depression scale (HADS). The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The anxiety and depression subscales each range from 0 to 21, with higher scores indicating higher anxiety/depression complains. Patients were defined as having anxiety or depression or both if the score was 8 or more in the corresponding subscale.
Change in dysfunctional breathing | Baseline - 24 weeks - 36 weeks
  This will be measured with the Nijmegen questionnaire. 16 questions will be asked, ranging from 0 to 4. The higher the score, the more likely it is that they have dysfunctional breathing.
Change in exercise capacity | Baseline - 24 weeks
  The functional exercise capacity will be measured by 6-minute walk test (6MWT).
Predictors of response in 6- minute walk distance (6MWD) | Post pulmonary rehabilitation
  The predictors will be based on baseline symptom scores (CAT, mMRC, CIS), baseline 6MWD and hospitalisation status.

OTHER OUTCOMES:
Evaluate the change in 6MWD after 6weeks or 12weeks PR. | Baseline - 6 weeks / 12 weeks
  The investigators will evaluate the 6MWD at 6 weeks and 12 weeks, as well as change in 6MWD from baseline to 6 weeks versus from baseline to 12 weeks PR.
Change in hand grip strength. | Baseline - 12 weeks
  This change will be objectived by measuring the hand grip strength with the Jamar hand-held dynamometer.
Change in respiratory muscle and diaphragm strength. | Baseline - 12 weeks
  This change will be objectived by measuring the maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP).
The cost-effectiveness of the intervention. | Baseline - end of the study
  In case the study findings on the primary outcome is positive, a cost-effectiveness analysis will be done to evaluate if the intervention had an impact on the health care costs verified through the financial expenses of patients.
Change in dyspnoea | Baseline - 12 weeks
  Changes in dyspnoea, measured with the modified medical research council (mMRC). The total mMRC scale ranges from 0 to 4 score where 0 represents no dyspnoea and 4 a lot of dyspnoea.
Change in sleep efficiency. | Baseline - 12 weeks
  The change in sleep efficiency will be measured by an activity tracker.
Change in functional status | Baseline - 12 weeks
  The functional status will be measured by the post COVID-19 functional status scale (PCFS). It is an ordinal score ranging from 0 to 4 where 4 means the patient has a lot of limitations in daily life.
Change in anxiety and depression symptoms. | Baseline - 12 weeks
  This will be measured by the Hospital Anxiety and depression scale (HADS). The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The anxiety and depression subscales each range from 0 to 21, with higher scores indicating higher anxiety/depression complains. Patients were defined as having anxiety or depression or both if the score was 8 or more in the corresponding subscale.
Change in work productivity and activity impairment. | Baseline - 12 weeks
  This will be measured with the "work productivity and activity impairment" questionnaire (WPAI), consisting of 6 questions.
Change in dysfunctional breathing | Baseline - 12 weeks
  This will be measured with the Nijmegen questionnaire. 16 questions will be asked, ranging from 0 to 4. The higher the score, the more likely it is that they have dysfunctional breathing.

CONTACTS AND LOCATIONS:
Overall Officials: Thérèse Lapperre, Prof., Principal Investigator — University Hospital, Antwerp
Locations (2):
- Belgium (2):
  - UHAntwerp, Edegem, Antwerp
  - Ziekenhuis Oost-Limburg, Genk, Limburg

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted starting after the publication of the primary endpoint and either publication of the follow-up data article or one year after the clinical study report is provided to the funder, whichever happens earlier. The data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to anonymized trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) by the TSC and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact purecovid@uza.be . An administrative cost may apply.

REFERENCES:
- [Derived] Volckaerts T, Ruttens D, Quadflieg K, Burtin C, Cops D, De Soomer K, Roelant E, Verhaegen I, Daenen M, Criel M, Vissers D, Lapperre T. Improved functional exercise capacity after primary care pulmonary rehabilitation in patients with long COVID (PuRe-COVID): a pragmatic randomised controlled trial. BMJ Open Respir Res. 2025 Nov 17;12(1):e003653. doi: 10.1136/bmjresp-2025-003653. PMID 41253410
- [Derived] Volckaerts T, Vissers D, Burtin C, Van Meerbeeck X, de Soomer K, Oostveen E, Claes K, Roelant E, Verhaegen I, Thomeer M, Criel M, Quadflieg K, Cops D, Ruttens D, Lapperre TS. Randomised, controlled, open-label pragmatic trial evaluating changes in functional exercise capacity after primary care PUlmonary REhabilitation in patients with long COVID: protocol of the PuRe-COVID trial in Belgium. BMJ Open. 2023 Jun 2;13(6):e071098. doi: 10.1136/bmjopen-2022-071098. PMID 37270195
- See also: Published PuRe-COVID protocol — https://bmjopen.bmj.com/content/13/6/e071098